CLINICAL TRIAL: NCT00348205
Title: A Study to Evaluate the Safety and Effectiveness of the Technols 217z Zyoptix System for Hyperopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 369
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Hyperopia; Astigmatism
MeSH Terms: conditions — Hyperopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Technolas 217z Zyoptix System (Experimental): Bausch & Lomb Technolas 217z Zyoptix System with Treatment Planner Customized Treatment Calculation Software.
  Interventions: Device: Technolas 217z Zyoptix Laser

INTERVENTIONS:
Device: Technolas 217z Zyoptix Laser — Technolas 217z Zyoptix System with Treatment Planner Customized Treatment Calculation Software for the wavefront-guided LASIK treatment of hyperopia and hyperoptic astigmatism.

SUMMARY:
A study to demonstrate the safety and effectiveness of wavefront laser refractive surgery treatments for hyperopia and astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Hyperopia with or without astigmatism.

Exclusion Criteria:

* Contraindications to LASIK.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-06; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Technolas 217z Zyoptix System
Started | 80
Completed | 78
Not Completed | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Zyoptix System
Number analyzed (Participants) | 80
Number analyzed (eyes) | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Uncorrected Visual Acuity (UCVA) of 20/40 or Better at 12 Months and 24 Months
Time Frame: 24 months
Population: The number of eyes available for uncorrected visual acuity assessment at 12 months and 24 months were included in the analysis.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Zyoptix System
Number analyzed (Participants) | 74
Number analyzed (eyes) | 147
eyes
  12 months | 147
  24 months: number analyzed (Participants) | 72
  24 months: number analyzed (eyes) | 143
  24 months | 140

2. Primary Outcome: Percentage of Eyes With a Postoperative Subjective Manifest Refraction Spherical Equivalent (MRSE) Within ± 1.00 Diopter (D) and ± 0.50 D of Emmetropia.
Description: Manifest refractions (eyeglass prescriptions) have three components: sphere, cylinder, and axis. Sphere and cylinder are both expressed in diopters, which is a continuous measure of the focusing power needed to make the image sharp on the retina. Manifest refraction spherical equivalent (MRSE) is equal to sphere + ½ x cylinder. It is expressed in diopters (D).
Time Frame: 12 months
Population: The number of eyes available for manifest refraction spherical equivalent assessment at 12 months were included in the analysis.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Zyoptix System
Number analyzed (Participants) | 74
Number analyzed (eyes) | 147
eyes
  Within 0.50 D | 100
  Within 1.00 D | 142

3. Primary Outcome: The Percentage of Eyes With a Postoperative Subjective Manifest Refraction Spherical Equivalent (MRSE) Within ± 1.00 Diopter (D) and ± 0.50 D of Emmetropia
Description: as for outcome 2
Time Frame: 24 months
Population: The number of eyes available for manifest refraction spherical equivalent assessment at 24 months were included in the analysis.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Zyoptix System
Number analyzed (Participants) | 72
Number analyzed (eyes) | 143
eyes
  Within 0.50 D | 97
  Within 1.00 D | 129

4. Primary Outcome: Refractive Stability - Categorical Change Between Month 1 and Month 3
Description: Percentage of eyes with a change of ≤ 1.00 Diopter in manifest refraction spherical equivalent (MRSE) between postoperative refractions, performed at 1 months and 3 months after surgery. Manifest refractions (eyeglass prescriptions) have three components: sphere, cylinder, and axis. Sphere and cylinder are both expressed in diopters, which is a continuous measure of the focusing power needed to make the image sharp on the retina. Manifest refraction spherical equivalent (MRSE) is equal to sphere + ½ x cylinder. It is expressed in diopters (D).
Time Frame: Month 1, Month 3
Population: There were 139 eyes with manifest refraction spherical equivalent assessments at both Month 1 and Month 3 for this outcome assessment.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Zyoptix System
Number analyzed (Participants) | 70
Number analyzed (eyes) | 139
eyes | 135

5. Primary Outcome: Refractive Stability - Mean Change Between Month 1 and Month 3
Description: Mean change in manifest refraction spherical equivalent (MRSE) between postoperative refractions, performed at 1 months and 3 months after surgery. Manifest refractions (eyeglass prescriptions) have three components: sphere, cylinder, and axis. Sphere and cylinder are both expressed in diopters, which is a continuous measure of the focusing power needed to make the image sharp on the retina. Manifest refraction spherical equivalent (MRSE) is equal to sphere + ½ x cylinder. It is expressed in diopters (D).
Time Frame: 1 month, 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Zyoptix System
Number analyzed (Participants) | 70
Number analyzed (eyes) | 139
diopter | 0.12 (0.40)

6. Primary Outcome: Induced Astigmatism
Description: Percentage of eyes which had >2.00 Diopter of induced refractive cylinder for those eyes treated for spherical hyperopia only.
Time Frame: 24 months
Population: There were 32 sphere eyes assessed for this outcome measure.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Zyoptix System
Number analyzed (Participants) | 16
Number analyzed (eyes) | 32
eyes | 0

7. Secondary Outcome: Loss of Best Spectacle-corrected Visual Acuity (BSCVA)
Description: Percentage of eyes with loss of best spectacle corrected visual acuity (BSCVA) of >2 lines. Mean change in best-corrected high contrast distance visual acuity. Corrected means spectacle corrected. Visual acuity (VA) was reported as letters read correctly, and the letters read were converted to logarithm of the minimum angle of resolution (logMAR) acuity. The participant read rows of letters on a standard LogMAR chart until the participant misses 3 letters on a row with 5 letters. The total number of correct letters were recorded. A decrease in the number of correct letters indicates a decrease in visual acuity. Acuity was averaged across visits.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Zyoptix System
Number analyzed (Participants) | 78
Number analyzed (eyes) | 155
eyes
  12 months | 1
  24 months: number analyzed (Participants) | 75
  24 months: number analyzed (eyes) | 150
  24 months | 3

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events (AEs) were assessed throughout the study. AEs were not coded (therefore, there is no source vocabulary).
Arm/Group | Technolas 217z Zyoptix System
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 1/80
Other Adverse Events (participants affected / at risk) | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Technolas 217z Zyoptix System (N=80)
Suction break (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.